CLINICAL TRIAL: NCT07222592
Title: MOBoxy: MoblO2 to Maintain Oxygenation
Acronym: MOBoxy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Stanford University (Other); Minnesota Health Solutions (Industry)
Responsible Party: Principal Investigator, Jeff Swigris, Professor of Medicine, National Jewish Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HS 4311; R44HL160356 (NIH)
Record Dates: First submitted 2025-10-20; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: COPD; Interstitial Lung Disease
Keywords: COPD; interstitial lung disease; pulmonary fibrosis; supplemental oxygen; symptoms; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoblO2 control (Experimental): MoblO2 control
  Interventions: Device: MoblO2 control
- MoblO2 no control (No Intervention)

INTERVENTIONS:
Device: MoblO2 control — For the study, participants will be provided compressed gas oxygen tanks. The MoblO2 device will be attached to one D tank, and the other will be in reserve for if/when the first tank runs out, in which case, the MoblO2 device will be removed from the empty tank, attached to the reserve tank for use, and the first tank will be filled from the concentrator and left in reserve. For the next two weeks, whenever patients exert, they will be asked to use the D tanks with the MoblO2 system supplied by the study. During one of the weeks (Week A), the MoblO2 device will be in place atop the D cylinder and will collect data but not control O2 flow. For the other week (Week B), the MoblO2 device will be in place atop the D cylinder and will collect data and control O2 flow.
  Arms: MoblO2 control

SUMMARY:
Many patients with chronic lung disease (e.g., chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD)) require supplemental oxygen (O2) at some point during their disease course. Practitioners prescribe O2 to patients with chronic lung disease in hopes of the following: 1) that it will limit desaturation events and combat breathlessness, thus preventing the frustratingly slow pace and numerous rest breaks patients are forced to adopt while doing even simple tasks; 2) that it will allow patients to be more active physically (perhaps increase their ability to exercise) and socially (perhaps leave the home more often); 3) that it will stave off putative complications of hypoxemia (e.g., cognitive dysfunction, pulmonary hypertension) and 4) that it will improve health-related quality of life (HRQL).

However, despite the rationale for O2, and prescribers' good intentions, patients generally view O2 with frustration and fear - it threatens their HRQL, which is already impaired by having a condition that imposes itself on every aspect of their lives. Nasal cannulas and delivery devices call unwanted attention to patients when they are out in public. O2 users feel stigmatized and are often viewed as "smokers who get what they deserve, even if they never smoked a day in their lives" - or as disabled, sick or even infectious. O2 steals patients' independence, forcing them to plan their lives around it. The anxiety that patients and their caregivers experience around running out of oxygen, or not getting enough, immobilizes them and restricts participation in activities outside of the home. O2 disrupts the home environment, adding stress, and creating a burden for patients' caregiver-loved-ones who are often saddled with the responsibility of ensuring adequate equipment and supply of O2, and O2 is a constant reminder to patients they are living with a condition that could shorten their lives.

O2 delivery equipment is typically heavy, unwieldy and intimidating. Different recommendations (e.g., insurance companies use 88% as a cut-off for SpO2, while many practitioners focus on 90%) make it confusing for patients, which almost certainly affects adherence. O2-requiringpatients are starving for things that can make their lives easier. An auto-adjusting O2 delivery device - one that automatically delivers the correct amount of O2 to maintain blood oxygen at desired, pre-set levels - would alleviate the need for patients to constantly (incessantly for many) monitor their peripheral oxygen saturation (SpO2) and adjust O2flow to meet the demands as exertion levels vary .

The MoblO2 device is a battery-operated, light-weight, closed-loop O2 delivery device that houses a regulator (which attaches to compressed gas O2 tanks) and adjusts O2 flow to meet a pre-set blood oxygen level. A pulse oximeter is worn on the ear and transmits via Bluetooth to the device, which adjusts an internal valve to control flow on a second-to-second basis.

The user sets the dial to the highest flow of O2 needed to meet the demands of activities they might perform (up to 15 liters per minute), and the device adjusts flow, up to the pre-set level to maintain SpO2 at a preset level (e.g., > 90%). To conserve O2 supply in the tank - and to avoid over-oxygenation (which could be problematic for a small percentage of patients with the most severe COPD) - the MoblO2 begins to limit O2 flow at a SpO2 of 93%. The device can be manually over-ridden by the user, and should the battery run out - or the device fail for some unforeseen reason - the default position is valve open, so the users receive whatever flow of oxygen has been set on the dial.

Given the substantial burdens of O2 on patients and their families, the hassles patients describe with having to monitor their SpO2 and repeatedly adjust the flow of O2 to meet their needs, patients and experts around the world have called for improvements in O2 delivery equipment. The MoblO2 is just such a remarkable improvement and a giant step forward in helping to ease the burdens of O2 on patients who require it.

The purpose of this study is to investigate the effects of the MoblO2 O2 delivery device on a range of outcomes, including physical activity, amount (liters) O2 use; maintenance of adequate SpO2 levels; patient reported outcomes including symptoms, HRQL and satisfaction with the MoblO2 O2 device.

DETAILED DESCRIPTION:
This is a two-center (National Jewish Health and Stanford University), three-week, unblinded (to O2 delivery), cross-over trial of the MoblO2 device in patients with COPD or ILD who do not require O2 at rest but have been prescribed O2 for use with activity.

Once enrolled, each subject will be given an activity monitor and wear it for one week while using their own O2 device as they normally would. After week one, they will continue to wear the activity monitor and be provided a home-fill, stationary O2 concentrator and two D tanks (cylinders) that they will fill from the concentrator. The MoblO2 device will be attached to one D tank, and the other will be in reserve for if/when the first tank runs out, in which case, the MoblO2 device will be removed from the empty tank, attached to the reserve tank for use, and the first tank will be filled from the concentrator and left in reserve.

For the next two weeks, whenever patients exert, they will be asked to use the D tanks with the MoblO2 system supplied by the study. During one of the weeks (Week A), the MoblO2 device will be in place atop the D cylinder and will collect data but not control O2 flow. For the other week (Week B), the MoblO2 device will be in place atop the D cylinder and will collect data and control O2 flow.

III.B.1. Screening to establish O2 flow: Consented patients will be screened for O2 needs via an O2 titration protocol as follows: patients will be instructed to walk as fast as possible (without running or jogging) back and forth on a 30-meter course in quiet, low-traffic hallway while their SpO2 is monitored. The walk continues until 3 minutes are completed or SpO2 falls to ≤ 88%. If SpO2 does not fall to ≤ 88% by 3 minutes, the patient does not qualify for the study. If SpO2 falls to ≤ 88% before 3 minutes, the walk is halted, and the patient rests for 5 minutes. O2 is then added in 2L/min increments - continuous flow O2, delivered via an E tank on a trolley that the patient pulls while walking - until the patient is able to complete 3 minutes without the SpO2 falling to ≤ 88% for 15 seconds or more. Five-minute rest periods will be ensured between all walks.

Patients who need > 15 L/min O2 will be excluded. Because patients may exert to degrees greater than they did during the screening walks, for the week of the study that the MoblO2 device is in control mode the flow set on the device will be the higher of the following: 1) the flow determined by the screening protocol or 2) the highest flow that a patient has used in the last week.

III.B.2. Randomization: Which of the two weeks (A or B) the MoblO2 device will control O2 flow will be randomly assigned via a random number generator; thus, subjects could be randomized to either order: AB or BA. Each of the two sites will randomly assign the order.

Patient subjects will have previously-diagnosed COPD or chronic ILD and will have been prescribed by their treating practitioner O2 for use with exertion (but not at rest) for at least one month prior to enrollment. In total, 48 subjects will be recruited: 24 from National Jewish Health and 24 from Stanford University. At each site, 12 subjects will have COPD, and 12 subjects will have ILD.

The study will include a number of assessment tools, including actigraphy and patient-reported outcome measures. The Actigraph used is the GT3X + Tri-Axis Actigraphy Monitor (Actigraph LLC; Pensacola, FL) worn on the waist using the provided manufacturer's bands. Subjects will be asked to wear the Actigraph during waking hours, except when bathing or showering. Subjects will receive a charger, and they will be asked to charge the device overnight. Actigraph proprietary software will be used to generate values for sedentary time and time spent in moderately vigorous physical activity.

All questionnaires will be administered in electronic format via REDcap and in the same order at each visit. For subjects with COPD, the order will be: CAT, O2 satisfaction survey, FSS, IPAQ, Proactive, PGI-Dyspnea, PGI-Cough, PGI-Energy, and PGI-QOL. For subjects with ILD, the order will be: L-PF, O2 satisfaction survey, FSS, IPAQ, Proactive, PGI-Dyspnea, PGI-Cough, PGI-Energy, and PGI-QOL.

Outcome analyses. The initial analyses will compare the MoblO2 controlling O2 flow vs. not. In other analyses, the investigators will compare the MoblO2 controlling O2 flow vs. baseline. The following outcomes will be analyzed using a generalized linear model, with the difference in outcome of interest as the dependent variable:

* Activity outcomes (time spent in moderately vigorous physical activity or sedentary time)
* Oxygen outcomes (total liters used, MoblO2 over-rides (per hour)
* Saturation outcomes (% time with SpO2 < 90%, % time with SpO2 < 88%, number of desaturation events < 88% per hour)
* Questionnaire outcomes (CAT score, L-PF scores (Symptoms Module, Dyspnea domain, Cough domain, Energy domain, Impacts Module, L-PF total), IPAQ, Proactive, FSS and PGI)
* Oxygen satisfaction survey

ELIGIBILITY:
Inclusion Criteria:

1. Previously-diagnosed COPD or chronic ILD
2. Prescribed O2 for use with exertion at least 1 month prior to enrollment
3. Age 25 years old or greater
4. Self-reported stable symptoms and stable oxygen needs for at least 2 weeks
5. Patient consent to using compressed gas tanks to deliver O2 during the 2-week study period.

Exclusion Criteria:

1. Active angina
2. Hemoglobin less than 10mg/dL
3. Musculoskeletal disease that precludes physical activity
4. Ongoing participation or plans for participation in pulmonary rehabilitation during the study
5. Need for O2 at rest
6. Patient needing more than 10 L/min continuous flow with exertion on O2 screen. Patient prescribed 10L/min continuous flow (or more) by their prescribing physician

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Moderately vigorous physical activity (MVPA) | 1 week with the MoblO2 controlling O2 flow and 1 week with MoblO2 not controlling O2 flow
  Time spent in moderately vigorous physical activity as assessed by actigraphy

SECONDARY OUTCOMES:
COPD Assessment Test | 1 week change from baseline for each arm
  Symptom assessment for patients with COPD. The total score ranges from 0 to 40, with higher scores suggesting a greater impact of COPD on a patient's health.
Living with Pulmonary Fibrosis (L-PF) questionnaire scores | 1 week change from baseline for each arm
  Disease specific questionnaire for patients with ILD. The L-PF is a 44-item questionnaire that yields six scores (Symptoms Module, Dyspnea domain, Cough domain, Energy domain, Impacts Module, and Total), each ranging from 0 to 100, with higher scores indicating worse symptoms or greater negative impact of disease.

OTHER OUTCOMES:
Oxygen use | 1 week change from baseline for each arm
  O2 use each week, MoblO2 over-rides per week
Saturation outcomes | 1 week change from baseline for each arm
  (Percent (%) time with SpO2 < 90%, % time with SpO2 < 88%, number of desaturation events < 88% per hour
Patient reported outcome measures | 1 week
  International Physical Activity Questionnaire (long form) asks respondents to state how much time they spent doing various activities over the last seven days.
Patient reported outcome measures | 1 week
  PROactive Physical Activity in COPD (C-PPAC) instrument combines 14 items to generate a score ranging from 0-64, with higher scores indicating better status.
Patient reported outcome measures | 1 week
  Fatigue Severity Scale (FSS) is a 9-item questionnaire that measures fatigue. Scores range from 0-63, with higher scores indicating greater fatigue.
Patient reported outcome measures | 1 week
  Patient global impressions includes three items assessing shortness of breath, quality of life, and energy. Scores range from 0-15, with higher scores indicating worse status.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Swigris, DO, MS, Principal Investigator — National Jewish Health
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study designed to begin the assessment process for the MoblO2 device.

REFERENCES:
- [Background] Lindell KO, Collins EG, Catanzarite L, Garvey CM, Hernandez C, Mclaughlin S, Schneidman AM, Meek PM, Jacobs SS. Equipment, access and worry about running short of oxygen: Key concerns in the ATS patient supplemental oxygen survey. Heart Lung. 2019 May-Jun;48(3):245-249. doi: 10.1016/j.hrtlng.2018.12.006. Epub 2018 Dec 28. No abstract available. PMID 30598231
- [Background] Cardenosa SC, Palomo M, Francesqui J, Alsina X, Hernandez C, Albacar N, Blanco I, Embid C, Barbera JA, Hernandez-Gonzalez F, Sellares J. Home Oxygen Monitoring in Patients with Interstitial Lung Disease. Ann Am Thorac Soc. 2022 Mar;19(3):493-497. doi: 10.1513/AnnalsATS.202103-319RL. No abstract available. PMID 34793688
- [Background] Swigris JJ. Transitions and touchpoints in idiopathic pulmonary fibrosis. BMJ Open Respir Res. 2018 Jun 29;5(1):e000317. doi: 10.1136/bmjresp-2018-000317. eCollection 2018. PMID 30018766
- [Background] Earnest MA. Explaining adherence to supplemental oxygen therapy: the patient's perspective. J Gen Intern Med. 2002 Oct;17(10):749-55. doi: 10.1046/j.1525-1497.2002.20218.x. PMID 12390550
- See also: Website for Live Fully, Inc., the company that owns the patent for and rights to the MoblO2 — https://www.livefullyinc.com/